CLINICAL TRIAL: NCT07314346
Title: A Phase 1, Open-Label, Two-Part, Single-Sequence Study to Evaluate the Effect of Multiple Oral Doses of BEM/RZR FDC on the Pharmacokinetics of Buprenorphine/Naloxone or Methadone in Participants on Stable Maintenance Therapy for Opiate Withdrawal
Brief Title: Drug-drug Interaction Study of Bemnifosbuvir/Ruzasvir (BEM/RZR) and Buprenorphine/Naloxone or Methadone
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Atea Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AT-01B-013
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteer Study
MeSH Terms: interventions — Buprenorphine; Naloxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- (n=16) buprenorphine/naloxone + BEM/RZR (Experimental)
  Interventions: Drug: Buprenorphine/Naloxone + BEM/RZR
- (n=16) methadone + BEM/RZR (Experimental)
  Interventions: Drug: Methadone +BEM/RZR

INTERVENTIONS:
Drug: Buprenorphine/Naloxone + BEM/RZR — Day -5 to Day -1:buprenorphine/naloxone as individualized QD doses up to 24mg/6mg.
  Day 1 to Day 5:Individualized QD doses of buprenorphine/naloxone. Day 6 to Day 12:Individualized QD doses of buprenorphine/naloxone + BEM 550mg/RZR 180mg QD.
  Day 13 Individualized QD doses of buprenorphine/naloxone.
  Other Names: BEM (AT-527)/RZR (AT-038)
  Arms: (n=16) buprenorphine/naloxone + BEM/RZR
Drug: Methadone +BEM/RZR — Day -5 to Day -1:methadone individualized QD doses: 30-150mg. Day 1 to Day 5:Individualized QD does of methadone. Day 6 to Day 12:Individualized QD doses of methadone + BEM 550mg/RZR 180mg QD. Day 13 Individualized QD doses of methadone.
  Other Names: BEM (AT-527)/RZR (AT-038)
  Arms: (n=16) methadone + BEM/RZR

SUMMARY:
Drug-drug interaction study between Bemnifosbuvir/Ruzasvir (BEM/RZR) and Buprenorphine/Naloxone or Methadone

ELIGIBILITY:
Inclusion Criteria:

* Must agree to use acceptable contraceptive methods through at least 90 days after the last dose of study drug.
* Minimum body weight of 50 kg and body mass index (BMI) of 18-32 kg/ m2.
* Willing to comply with the study requirements and to provide written informed consent.

Exclusion Criteria:

* Infected with hepatitis B virus, hepatitis C virus, HIV.
* Abuse of alcohol or drugs.
* Use of other investigational drugs within 28 days prior to Day -5.
* Concomitant use of prescription medications, or systemic over-the-counter medications (apart from methadone or buprenorphine/naloxone as assigned maintenance therapy).
* Other clinically significant medical conditions or laboratory abnormalities.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-05-29 (Estimated); Study Completion 2026-05-29 (Estimated)

PRIMARY OUTCOMES:
Effect of BEM/RZR on PK of buprenorphine,norbuprenorphine and naloxone | Day -5 to Day 13
  Cmax
Effect of BEM/RZR on PK of buprenorphine,norbuprenorphine and naloxone | Day -5 to Day 13
  AUC
Effect of BEM/RZR on PK of methadone | Day -5 to Day 13
  Cmax
Effect of BEM/RZR on PK of methadone | Day -5 to Day 13
  AUC

CONTACTS AND LOCATIONS:
Locations (1):
- Atea Study Site, Overland Park, Kansas, United States